CLINICAL TRIAL: NCT06523439
Title: Investigating a Truncated Version of SAINT in Treatment-Naive Adolescents With Depression: An Open-Label Acceptability Trial
Brief Title: Accelerated Intermittent Theta Burst in Treatment-Naive Adolescents
Acronym: SAINT-KID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Magnus Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NECMHR01-FY24-032
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder; Depression in Adolescence; Depression; Major Depressive Episode
Keywords: Stanford Accelerated Intelligent Neuromodulation Therapy; SAINT; Transcranial Magnetic Stimulation; Accelerated Theta Burst Stimulation; Accelerated Intermittent Theta Burst Stimulation; TMS; TMS in Adolescents
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Single-blinded
Who Masked: Outcomes Assessor
Masking Description: Raters will be blinded as to whether the adolescent participants received Standard SAINT® (10 TMS treatments per day for 5 days) or Truncated SAINT® (5 TMS treatments per day for 5 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard SAINT® (Active Comparator): 10 daily sessions (50 total over 5-days) of SAINT® stimulation (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds), delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex).
  Interventions: Device: MagPro X100 edition (MagVenture, Skovlunde, Denmark)
- Truncated SAINT® (Experimental): 5 daily sessions (25 total over 5-days) of SAINT® stimulation (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds), delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex).
  Interventions: Device: MagPro X100 edition (MagVenture, Skovlunde, Denmark)

INTERVENTIONS:
Device: MagPro X100 edition (MagVenture, Skovlunde, Denmark) — 10 daily sessions (50 total over 5-days) of SAINT® (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds) guided by MNS, delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex).
  Other Names: Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT®) with Magnus Neuromodulation System (MNS)
  Arms: Standard SAINT®
Device: MagPro X100 edition (MagVenture, Skovlunde, Denmark) — 5 daily sessions (25 total over 5-days) of SAINT® (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds) guided by MNS, delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex).
  Other Names: Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT®) with Magnus Neuromodulation System (MNS)
  Arms: Truncated SAINT®

SUMMARY:
This is a single-site open-label clinical trial of the Stanford Accelerated Intermittent Neuromodulation Therapy (SAINT®) protocol. The goal of this clinical trial is to learn if a new form of transcranial magnetic stimulation (TMS)-known generally as accelerated intermittent theta burst stimulation (aiTBS) and specifically as SAINT®-is effective as a first-line therapy in treating adolescents aged 14-19 years-old in their first episode of depression who have not undergone a full course of depression treatment prior to starting the trial and who remain antidepressant-free throughout the trial.

The main questions this trial aims to answer are:

* Does SAINT® relieve symptoms of depression as a first-line therapy in adolescents?
* Is SAINT® a feasible option as a first-line treatment for adolescent depression?

Researchers will measure the depression symptoms in adolescent participants before and after SAINT®. Parents of the adolescent participant will also participate in the study providing information about their experience and preference for TMS as a first-line treatment.

Adolescent participants will:

* Remain antidepressant-free throughout the study period of 6-7 weeks.
* Receive an MRI of their head for precision targeting
* Receive 5 days of aiTBS (SAINT®)

DETAILED DESCRIPTION:
This single-site open-label clinical trial aims to test the safety and efficacy of the Magnus Neuromodulation System (MNS) with Stanford Accelerated Intermittent Neuromodulation Therapy (SAINT®) technology in treatment-naive adolescents with major depressive disorder (MDD) who remain antidepressant-free throughout the treatment. The SAINT® protocol, or a truncated version (5 or 10 applications per day to a customized target within the left dorsolateral prefrontal cortex [L-DLPFC] identified with fMRI for five consecutive days), in combination with MNS software will be delivered to each adolescent participant. Changes in depressive symptoms will be measured at baseline and two follow up visits. Additionally, parents and adolescents will answer questions regarding their preference for SAINT® as a first-line treatment option for MDD.

The hypothesis is that adolescent participants receiving SAINT® or the truncated version will demonstrate similar response and remission rates that are comparable to SAINT® trials in adults (80-90%) as measured by the Childhood Depression Rating Scale (CDRS) and Hamilton Depression Rating Scale.

The primary objective of this study is to determine the efficacy of active SAINT® in reducing symptoms of depression as measured by the CDRS at the one-month follow up time point.

The study will enroll approximately 40 participants and employ a two-arm design with 20 participants per arm. The target population is adolescents of all genders and ethnicities who are between 14 and 19 years of age with a diagnosis of MDD experiencing their first major depressive episode who have not received a full course of prior treatment and who are otherwise in good general health. Participants must be without contraindications to Magnetic Resonance Imaging (MRI) or transcranial magnetic stimulation (TMS) and must be able to attend all study visits.

This study will deliver SAINT® via a MagPro X100 edition (MagVenture, Skovlunde, Denmark) TMS device equipped with a Cool-B65 A/P coil. The stimulation paradigm consists of 5 or 10 daily sessions (25 or 50 total over 5-days) of SAINT® (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds) guided by MNS, delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, between the ages of 14 and 19 at the time of screening.
2. Able to read, understand, and provide written, dated assent and/or consent prior to screening. Proficiency in English sufficient to complete questionnaires and follow instructions during aiTBS interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
3. Diagnosed with Major Depressive Disorder (MDD) with a current Major Depressive Episode (MDE), according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
4. No prior major depressive episodes (MDEs) as determined by MINI-KID
5. HAMD-17 score of ≥20 at screening (Visit 1).
6. Treatment-naive as determined by the ATHF (no adequate antidepressant trials prior to screening defined as fewer than 4 weeks of antidepressant medication and fewer than 8 psychotherapy sessions in lifetime; willingness to taper medications and stop psychotherapy if recently started and within the window defined above.)
7. TMS naive.
8. Access to ongoing psychiatric care before and after completion of the study.
9. In good general health, as evidenced by medical history.
10. Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

1. Pregnancy
2. High-risk for suicide or active suicidal ideation (Suicidal Ideation Questionnaire- Junior [SIQ-JR] ≥ 31).
3. The presence or diagnosis of prominent anxiety disorder, or dysthymia (>3 on SAPAS; >10 on GAD-7)
4. Current severe insomnia (must sleep a minimum of 5 hours each night before stimulation)
5. Current mania or psychosis
6. Bipolar Affective Disorder and/or primary psychotic disorders.
7. Autism Spectrum disorder or Intellectual Disability
8. A diagnosis of obsessive-compulsive disorder (OCD)
9. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal.
10. Urine screening test positive for illicit substances.
11. Any history of ECT (greater than 8 sessions) without meeting responder criteria
12. Recent (during the current depressive episode) or concurrent use of a rapid acting antidepressant agent (i.e., ketamine or a course of ECT).
13. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma.
14. Untreated or insufficiently treated endocrine disorder.
15. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
16. Contraindications to MRI (ferromagnetic metal in their body).
17. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
18. Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO)
19. Treatment with another investigational drug or other intervention within the study period.
20. Any other condition deemed by the PI to interfere with the study or increase risk to the participant.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Childhood Depression Rating Scale-Revised (CDRS-R) Remission Rates | Baseline, One Month Follow Up Visit
  Seventeen item diagnostic questionnaire which psychiatrists use to measure the severity of depressive symptoms in adolescents with depression.
  The investigators will assess the difference in CDRS-R scores/remission rates between Standard SAINT® group compared to those who received Truncated SAINT® at the one-month follow up visit.
Childhood Depression Rating Scale-Revised (CDRS-R) Remission Rates | Baseline, One Month Follow Up Visit
  The investigators will assess the difference in CDRS-R response rates (reduction >50% of CDRS-R baseline score) between the Standard SAINT® group compared to those who received Truncated SAINT®.

CONTACTS AND LOCATIONS:
Overall Officials: Sean J O'Sullivan, M.D., Ph. D., Principal Investigator — University of Texas at Austin
Locations (1):
- Dell Medical School at University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No